CLINICAL TRIAL: NCT01810627
Title: Application of Megavoltage Imaging to Reduce Artifact Following Interstitial Seed Implants for Prostate Adenocarcinoma
Brief Title: Application of Megavoltage Imaging to Reduce Artifact After Seed Implants
Status: Completed | Type: Observational
Sponsor: William St Clair (Other)
Responsible Party: Sponsor-Investigator, William St Clair, Faculty, Radiation Medicine, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 13-RAD-01
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MVCT: Patients will receive an additional MVCT scan at their one month follow up visit.
  Interventions: Radiation: MVCT

INTERVENTIONS:
Radiation: MVCT — Patients will receive an additional MVCT scan at their one month follow up visit.

SUMMARY:
This is a non-randomized study to evaluate the utility of MVCT as a quality assurance measure in patients treated with interstitial permanent seed implants for low and intermediate risk prostate cancer. All patients will received the same standard of care treatment but will receive an additinoal CT image of the prostate.

ELIGIBILITY:
Inclusion Criteria:

Male 50-80 years of age Eligible for interstitial brachytherapy implants

Exclusion Criteria:

-

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in prostate volume measured in cm^3 | One month post implant
  Change in prostate volume measured with trans-rectal ultrasound at baseline versus prostate volume measured with KVCT and MVCT.

CONTACTS AND LOCATIONS:
Overall Officials: William St. Clair, MD, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- Markey Cancer Center, Lexington, Kentucky, United States